CLINICAL TRIAL: NCT02569164
Title: Urinary Albumin Excretion in Women With Polycyclic Ovary Syndrome and it's Relation to Cardiovascular Risk Factors
Brief Title: Cardiovascular Risks and Urinary Albumin Excretion(UAE) in Polycystic Ovarian Syndrome (PCO)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, suzy abdelaziz Abdelhamid, lecturer of Obgyn, Kasr El Aini Hospital
Other Study IDs: kasrelaini Obgyn..
Record Dates: First submitted 2015-08-26; First posted 2015-10-06 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Urinary Albumin Excretion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
PCO patients will be assessed clinically,urine & blood samples will be tested. Systolic & diastolic blood pressure, serum glucose & insulin levels, lipid profile, C-reactive protein, complete hormonal profile, and Urinary albumin excretion will be measured.

DETAILED DESCRIPTION:
PCO patients with 2 of 3 criteria: oligo- or anovulation ; hyperandrogenism &polycystic ovaries. Exclusion criteria: pregnancy, diabetes, hypertension , adrenal & thyroid dysfunction.

Blood samples after overnight fast (8hrs) at day 2 or 3 of menstrual cycle. Serum concentration of follicle stimulating hormone (FSH), luteinizing hormone (LH), prolactin, total testosterone & sex hormone binding globulin, serum 17-hydroxy (OH) progesterone & dehydroepiandrosterone sulfate will be measured.

Oral glucose tolerance test & plasma insulin levels will be measured. Total cholesterol, triglycerides, high& low density lipoproteins. Urinary albumin will be measured& all the data will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* PCO patients

Exclusion Criteria:

* pregnancy
* diabetes
* hypertension
* adrenal dysfunction
* thyroid dysfunction

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: PCO patients
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-10; Primary Completion 2015-11 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with hyperinsulinemia (uIU/ml) | 3 months
Number of patients with hyperlipidemia (mg/dl). | 3 months
Number of patients with albuminuria(ug/ml) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: suzy abdelaziz, M.D., Principal Investigator — kasrelaini